CLINICAL TRIAL: NCT00753259
Title: The Effect of a Nurse-driven ICT-supported Disease Management Program to Improve the Treatment of Patients With Atrial Fibrillation.
Brief Title: Atrial Fibrillation (AF) Clinic to Improve the Treatment of Patients With Atrial Fibrillation.
Acronym: AFClinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Dr RG Tieleman, MD, PhD, Dept of Cardiology, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC 06-4-043
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-04

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; disease management program; integrated chronic care program; guideline; stroke; heart failure; quality of life; costs
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AF Clinic (Experimental)
  Interventions: Other: AF Clinic
- Care as Usual (Active Comparator)
  Interventions: Other: Care as Usual

INTERVENTIONS:
Other: AF Clinic — Treatment of atrial fibrillation patients by specialized nurses, supervised by cardiologists, using dedicated software to ensure maximal adherence to AHA/ACC/ESC guidelines on atrial fibrillation treatment
  Arms: AF Clinic
Other: Care as Usual — Routine clinical care of atrial fibrillation patients, provided by cardiologists, without the help of specialized nurses or dedicated software.
  Arms: Care as Usual

SUMMARY:
* Randomized controlled trial comparing specialized AF Clinic with 'care as usual'
* Hypothesis: treatment of AF patients in the AF-Clinic by a nurse, specialised in AF, using guideline-based dedicated software, under supervision of a cardiologist, is efficient, safe and not inferior to care as usual by a cardiologists.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed atrial fibrillation

Exclusion Criteria:

* Age < 18 years
* unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2006-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Composite of heart failure, thromboembolic complications, bleeding, severe adverse effects of drugs and death from cardiovascular causes. | minimum of 1 year

SECONDARY OUTCOMES:
All cause mortality, all cause hospitalizations, Treatment (benchmarking) in accordance to the 2006 AHA/ACC/ESC guidelines in AF, quality of life, patient satisfaction, anxiety, depression, compliance and cost effectiveness. | minimum of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Tieleman, MD PhD, Principal Investigator — Maastricht UMC
Locations (2):
- Netherlands (2):
  - Martini Hospital Groningen, Groningen
  - MaastrichtUMC, Maastricht

REFERENCES:
- [Derived] Hendriks JM, Vrijhoef HJ, Crijns HJ, Brunner-La Rocca HP. The effect of a nurse-led integrated chronic care approach on quality of life in patients with atrial fibrillation. Europace. 2014 Apr;16(4):491-9. doi: 10.1093/europace/eut286. Epub 2013 Sep 20. PMID 24058179
- [Derived] Hendriks JM, Crijns HJ, Tieleman RG, Vrijhoef HJ. The atrial fibrillation knowledge scale: development, validation and results. Int J Cardiol. 2013 Sep 30;168(2):1422-8. doi: 10.1016/j.ijcard.2012.12.047. Epub 2013 Jan 8. PMID 23305860
- [Derived] Hendriks JM, de Wit R, Crijns HJ, Vrijhoef HJ, Prins MH, Pisters R, Pison LA, Blaauw Y, Tieleman RG. Nurse-led care vs. usual care for patients with atrial fibrillation: results of a randomized trial of integrated chronic care vs. routine clinical care in ambulatory patients with atrial fibrillation. Eur Heart J. 2012 Nov;33(21):2692-9. doi: 10.1093/eurheartj/ehs071. Epub 2012 Mar 27. PMID 22453654
- [Derived] Hendriks JM, de Wit R, Vrijhoef HJ, Tieleman RG, Crijns HJ. An integrated chronic care program for patients with atrial fibrillation: study protocol and methodology for an ongoing prospective randomised controlled trial. Int J Nurs Stud. 2010 Oct;47(10):1310-6. doi: 10.1016/j.ijnurstu.2009.12.017. Epub 2010 Jan 20. PMID 20089253